CLINICAL TRIAL: NCT05936554
Title: Whole Body Vibration Versus Functional Strength Training On Balance In Children With Hemiparetic Cerebral Palsy: Randomized Comparative Study
Brief Title: Whole Body Vibration Versus Functional Strength Training On Balance In Children With Hemiparetic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amany Ibrahim AbdElhamed Sabra (Other)
Responsible Party: Sponsor-Investigator, Amany Ibrahim AbdElhamed Sabra, Bachelor's Degree of physical therapy, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EG, KFS lab Research
Record Dates: First submitted 2023-06-24; First posted 2023-07-07 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy; Hemiparesis
Keywords: cerebral palsy; Hemiparesis; balance; whole body vibration; functional strength training
MeSH Terms: conditions — Cerebral Palsy; Paresis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration (Active Comparator): will receive whole body Vibration training that elicits a warm up effect to improves muscle power and balance in addition to designed physical program.
  Interventions: Device: whole body vibration
- Functional strength training (Active Comparator): will receive Functional strength training that focuses on the movement pattern quality and treats functional movement and provides postural stability while promoting balance independence with confidence
  Interventions: Other: Functional strength training

INTERVENTIONS:
Device: whole body vibration — to improve muscle power and balance.
  Arms: whole body vibration
Other: Functional strength training — used in treatment of hemiparetic cerebral palsy and provides postural stability while promoting balance independence with confidence and muscle power
  Arms: Functional strength training

SUMMARY:
The study will be directed to compare which of whole body vibration (WBV) training and Functional strength training (FST) has better effect on balance in children with hemiparesis

DETAILED DESCRIPTION:
Hemiparesis is a type of hemiplegia where mild muscle weakness causes balance disturbances because one side of the body is affected such as the arm, chest leg or face.

Muscle weakness is commonly associated with abnormal bone development, leading to increased susceptibility to fractures, most cerebral palsy children have deficits in balance, coordination, and gait throughout childhood and adulthood. So, it is essential to seek an ideal physical therapy program to help in solving such widespread problem.

Balance control is important for competence in the performance of most functional skills, helping children to recover from unexpected balance disturbances, either due to slips and trips or to self- induced instability when making a movement that brings them toward the edge of their limit of stability Whole body vibration is mechanical oscillation, defined by amplitude and frequency, generates a force that acts on whole body. It is a training method for muscle tone modulation that is increasingly used in a variety of clinical situations.

Functional strength training (FST) is an effective method of exercise therapy. It can be combined with traditional physical therapy methods and can be successfully combined with most rehabilitation and exercise equipment. It provides postural stability while promoting independence with confidence.

The current study will be directed to compare which of whole body vibration (WBV) training and Functional strength training (FST) has better effect on balance in children with hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* The children in the study will be selected according to the following criteria:

  1. Their chronological age ranged from five to eight years old.
  2. Spasticity Grade I and II according to Modified Ashworth Scale.
  3. They will be on Level II and III according to Gross Motor Functional Classification System (GMFCS)
  4. Have the ability to walk independently.
  5. They can understand order and follow instruction.
  6. The child will be able to follow verbal commands and instructions.
  7. They can firmly grasp the rails of biodex device.

Exclusion Criteria:

1. Children with visual or auditory problems.
2. Children with uncontrolled convulsions.
3. Children with fixed contractures and deformities.
4. Children with surgical intervention less than one year.
5. Children injected by BOTOX in the calf muscle from less than one year.
6. Children had heart disease.
7. Children with epilepsy.
8. Children with severe diabetes.
9. Children with severe vascular disease

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-07-08 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Estimated)

PRIMARY OUTCOMES:
balance improvement | 3 months
  we will use pediatric balance scale and Biodex balance system to measure balance

SECONDARY OUTCOMES:
gross motor performance | 3 months
  we will use Gross Motor Function Measure 88 (GMFM-88) to measure gross motor performance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
For assessment :
  Modified Ashworth scale, Gross Motor Function Classification System Expanded and Revised (GMFCS-ER), The six-minute walk test (6MWT), Biodex stability system and pediatric balance scale.
  For Treatment:
  At first both groups will receive 60 minutes of designed physical therapy program, which consisted of stretching for the lower extremity muscles, namely hip flexors and adductors, hamstrings, and calf muscles: kneeling exercises, and standing and gait training as warming up then group I will receive whole body vibration (WBV) for 25 minutes and group II will receive functional strength training program (FST) for 30 minutes